CLINICAL TRIAL: NCT06887400
Title: Comparison of the Effectiveness of Focused Point-of-Care Ultrasonography Triage and Classical Triage in Patients Applying to the Emergency Department with Abdominal Pain
Brief Title: Pocus Triage in Patients Presenting to the Emergency Department with Abdominal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Necip Gökhan Güner, Assistant Professor,MD, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 16214662-050.01.04-319685-197
Record Dates: First submitted 2025-02-28; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Pain (AP); Point of Care Ultrasound (POCUS); Triage
Keywords: Emergency department; Abdominal pain; POCUS; Triage
MeSH Terms: conditions — Abdominal Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POCUS Triage (Experimental): Patients are directed to the area where they will be examined in accordance with the triage category determined by abdominal POCUS, which is performed in addition to classical triage.
  Interventions: Other: Point of care ultrasound (POCUS)
- Classical Triage (No Intervention): Patients are directed to the area where they will be examined in accordance with the triage category determined by classical triage application.

INTERVENTIONS:
Other: Point of care ultrasound (POCUS) — In this study, POCUS was performed by the same emergency medicine physician who had basic and advanced USG training and at least two years of POCUS experience, in accordance with ACEP imaging protocols. A portable USG device with B-Mode, M-Mode, Color Doppler, Power Doppler, Pulsed Wave Doppler modes, and which can be used in all clinical modes with a single probe was used during the protocol application (Butterfly iQ+™, Burlington, United States). Eight abdominal points (epigastric region, right upper quadrant, right side, right lower quadrant, suprapubic region, left lower quadrant, left side and upper quadrant, umbilical region) were scanned with POCUS, the findings were recorded on the previously prepared form, the triage categories of the patients (cl) were updated and the patients were directed to the area where they would be examined with the form.
  Arms: POCUS Triage

SUMMARY:
Introduction and Objective: This study aimed to reveal the effect of classical triage and Bedside Focused Ultrasonography (POCUS) in addition to classical triage on diagnosis, treatment, emergency department follow-up and its relationship with triage models in patients presenting to the emergency department with abdominal pain complaints.

METHOD: This randomized, controlled, prospective study was conducted with a total of 262 volunteer participants who were divided into two groups as 127 classical triage and 135 POCUS in addition to classical triage with non-traumatic abdominal pain. The decision of which participant would be included in which group was made at a 1:1 ratio using a computer-aided randomization table. The researcher did not intervene in the clinical processes in any way. In this study, the effect of POCUS application performed in addition to classical triage on clinical processes (imaging request, initial analgesia administration time, consultation request, emergency department stay and outcome) in the primary outcome and on triage systems in the secondary outcome were evaluated. IBM SPSS 21.0 software was used for statistical analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Present to the emergency room with abdominal pain
* No history of trauma in the last 48 hours
* Stable hemodynamics

Exclusion Criteria:

* According to the 3-way triage, the color code is red
* Being under the age of 18
* Being pregnant
* Having a history of trauma within the last 48 hours
* Being morbidly obese
* Having mental retardation
* Having repeated emergency room visits
* Being referred from the polyclinic to the emergency room with a diagnosis
* Filling the study form incompletely

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Time to initial analgesia | 6 months
  To evaluate the effect of adding the POCUS application to conventional triage on clinical processes, including imaging requests, time to initial analgesia.
Request for additional medical imaging | 6 months
  To evaluate the effect of adding the POCUS application to conventional triage on imaging requests.
Emergency department length of stay | 6 months
  To evaluate the effect of adding POCUS to conventional triage on the length of stay of patients in the emergency department.

OTHER OUTCOMES:
POCUS diagnostic sensitivity | 6 months
  To determine the diagnostic sensitivity of POCUS performed during triage using the final reports of patients who requested imaging.
Emergency severity index Outcome Measure | 6 months
  To examine the categorization changes after POCUS with the emergency severity index before POCUS application.
Manchester Triage System Outcome Measure | 6 months
  To examine the categorization changes after POCUS with Manchester triage system before POCUS application.
3-group triage system Outcome Measure | 6 months
  To examine the categorization changes after POCUS with 3-group triage system before POCUS application

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Training and Research Hospital, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thamburaj R, Sivitz A. Does the use of bedside pelvic ultrasound decrease length of stay in the emergency department? Pediatr Emerg Care. 2013 Jan;29(1):67-70. doi: 10.1097/PEC.0b013e31827b53f9. PMID 23283267
- [Background] Guner NG, Yurumez Y, Yucel M, Alacam M, Guner ST, Ercan B. Effects of Point-of-care Ultrasonography on the Diagnostic Process of Patients Admitted to the Emergency Department with Chest Pain: A Randomised Controlled Trial. J Coll Physicians Surg Pak. 2020 Dec;30(12):1262-1268. doi: 10.29271/jcpsp.2020.12.1262. PMID 33397050
- [Background] Durgun Y, Yurumez Y, Guner NG, Aslan N, Durmus E, Kahraman Y. Abdominal Pain Management and Point-of-care Ultrasound in the Emergency Department: A Randomised, Prospective, Controlled Study. J Coll Physicians Surg Pak. 2022 Oct;32(10):1260-1265. doi: 10.29271/jcpsp.2022.10.1260. PMID 36205268